CLINICAL TRIAL: NCT02241434
Title: The Role of Autologous Bone Marrow Mononuclear Cell Therapy in Duchenne Muscular Dystrophy
Brief Title: Stem Cell Therapy in Duchenne Muscular Dystrophy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-13
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; Autologous Bone marrow Mononuclear cell therapy; Stem Cells
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell (Experimental): bone marrow mononuclear cell transplantation
  Interventions: Biological: Stem Cell

INTERVENTIONS:
Biological: Stem Cell — Intrathecal autologous bone marrow mononuclear cell transplantation

SUMMARY:
The purpose of this study was to study the effect of stem cell therapy in patients with Duchenne Muscular Dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* age group of 3-25 years
* Duchenne muscular dystrophy diagnosed on the basis of clinical presentation

Exclusion Criteria:

* presence of respiratory distress
* presence of acute infections such as Human Immunodeficient Virus/Hepatitis B Virus/Hepatitis C Virus
* malignancies
* acute medical conditions such as respiratory infection, fever, hemoglobin less than 8, bleeding tendency, bone marrow disorder, left ventricular ejection fraction < 30%
* pregnancy or breastfeeding

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Manual Muscle Testing | 1 year

SECONDARY OUTCOMES:
Brooke and Vignos Scale | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Neurogen brain and spine institute, Navi Mumbai, Maharashtra, India